CLINICAL TRIAL: NCT05004675
Title: Randomized Open Label, Phase 3 Study to Compare the Efficacy and Safety of Lerodalcibep (LIB003) to Inclisiran in Patients at Very High or High Risk for CVD, on Stable Lipid-Lowering Therapy Requiring Additional LDL-C Reduction
Brief Title: Trial to Evaluate Efficacy and Safety of LIB003 and Inclisiran in High-risk CVD Patients
Acronym: LIBerate-VI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIB003-012
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Hypercholesterolemia; Atherosclerotic Ischemic Disease
Keywords: lerodalcibep; PCSK9 inhibitor; inclisiran
MeSH Terms: conditions — Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Intervention Model Description: randomized, comparative trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: efficacy parameters (lipids) blinded after randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- lerodalcibep (Experimental): 300 mg SC dosed monthly
  Interventions: Biological: lerodalcibep
- inclisiran (Active Comparator): 284 mg SC dosed Day 1 and Day 90
  Interventions: Drug: Inclisiran

INTERVENTIONS:
Biological: lerodalcibep — 300 mg
  Other Names: LIB003
  Arms: lerodalcibep
Drug: Inclisiran — 284 mg
  Other Names: Leqvio
  Arms: inclisiran

SUMMARY:
Comparison of LDL-C reductions of lerodalcibep (LIB003) 300 mg to inclisiran (Leqvio®) 284 in patients at very-high risk or high-risk for CVD on stable diet and oral LDL-C-lowering drug therapy

DETAILED DESCRIPTION:
Randomized, Open Label (lipids blinded), Phase 3 Study to Evaluate the Efficacy and Safety of Lerodalcibep (LIB003) at Day 270 of subcutaneous (SC) monthly (QM [≤31 days]) lerodalcibep (LIB003) 300 mg administered to SC inclisiran (Leqvio®) 284 mg at Days 1 and 90 in patients with very-high risk or high-risk CVD or at high risk for CVD with LDL-C ≥85 mg/dL on a stable diet and oral LDL-C-lowering drug therapy

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study-specific procedure;
* Weight of ≥40 kg (88 lb) and body mass index (BMI) ≥16 and ≤42 kg/m2;
* Very- high or high risk for CVD as defined in 2019 ESC/EAS Guidelines
* High-intensity statin (daily atorvastatin 40/80 or rosuvastatin 20/40) without other acceptable oral lipid lowering treatment plus diet; stable >4 weeks with LDL-C ≥85 mg/dL and triglycerides ≤400 mg/dL
* Women of childbearing potential (WOCBP) must continue using a highly effective form of birth control if sexually active
* Males whose partners are of CBP and not using a highly effective form of birth control will either be surgically sterile or agree to use the following forms of contraception, male or female condom with spermicide

Exclusion Criteria:

* Prior or active clinical condition or acute and/or unstable systemic disease, including cancer, compromising patient inclusion or preclude completion of the study, at the discretion of the Investigator
* Homozygous FH
* non-high intensity statins, mipomersen, lomitapide, gemfibrozil, and bempedoic acid
* PCSK9 mAb within 4 weeks of screening or siRNA within 1 year
* Severe renal dysfunction, defined eGFR <30 ml/min
* Recent, within 3 months of screening, atherosclerotic event or intervention
* planned cardiac procedure
* NYHA class III or IV heart failure
* active liver disease
* uncontrolled diabetes defined as fasting glucose >200 mg/dL and HbA1c > 9%
* uncontrolled BP ≥180 mmHg systolic or ≥110 mmHg diastolic;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
LDL-C change | Day 270
  Percent LDL-C change from baseline

SECONDARY OUTCOMES:
Adverse Events | 270 days
  frequency and severity of injection site reactions (ISRs)
Serum free PCSK9 levels | Day 270
  Percent change in free PCSK9 from baseline
Apolipoproteins | Day 270
  Percent change in Apo B and Lp(a) from baseline
Treatment goal achievement | Day 270
  Percent of patients reaching ESC/EAS treatment goals

CONTACTS AND LOCATIONS:
Overall Officials: Evan A Stein, MD PhD, Study Director — LIB Therapeutics
Locations (7):
- France (2):
  - CHU de Nantes - Hôpital Nord Laennec, Nantes, Cedex 01
  - Hopitaux de Marseille, Marseille, Cedex 05
- Universitätsklinikum Heidelberg - Medizinische Klinik, Heidelberg, Germany
- The Lipid Clinic (Oslo University Hospital), Oslo, Nydalen, Norway
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- United Kingdom (2):
  - Oak Tree Surgery and Pensilva Health Centre, Liskeard, Cornwall
  - Ashton Medical Group, Ashton-under-Lyne, Lancashire

IPD SHARING:
Plan to Share IPD: No